CLINICAL TRIAL: NCT01327430
Title: Effect of a Milk Phospholipid Supplementation on the Lipid Metabolism in Healthy Volunteers
Brief Title: Phospholipid Absorption of a Milk Phospholipid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Prof. Dr. G. Jahreis, Friedrich Schiller University of Jena, Department of Nutritional Physiology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LSEP H44-10
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: glycerophosphates; sphingomyelins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phospholipid supplementation (Experimental): Supplementation of milk phospholipid
  Interventions: Dietary Supplement: Milk phospholipid

INTERVENTIONS:
Dietary Supplement: Milk phospholipid — During day 1 until 10 the subjects were supplemented with daily 3 g milk phospholipids, during the day 11 and 20 the supplementation was increased to daily 6 g, and during the day 21 and 30 the subjects received daily 6 g milk phospholipids and 2 g of plant sterols.

SUMMARY:
The aim of the study is to investigate parameters of the lipid metabolism in plasma and feces of healthy subjects after a dietary supplementation of different dosages of milk phospholipids.

DETAILED DESCRIPTION:
To date the mechanisms for the intestinal absorption of glycerophosphates and sphingolipids are not completely investigated. It is assumed, that sphingolipids and sterols compete for intestinal absorption. In addition it is unclear, if a dietary phospholipid supplementation may influence the phospholipid concentration in plasma.

To evaluate the effect of a dietary phospholipid supplementation 15 healthy female subjects received over 10 days daily 3 g of milk phospholipids stirred in a dairy product. During the following 10 days the subjects were supplemented with daily 6 g milk phospholipid. Finally, the subjects received over 10 days 6 g of the milk phospholipid in a dairy product and 2 g of plant sterols serving a commercial product.

ELIGIBILITY:
Inclusion Criteria:

* female
* age: between 30 and 45 years

Exclusion Criteria:

* metabolic diseases
* arteriosclerosis
* pregnancy and breast feeding

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in plasma phospholipid concentration | after 0, 10, 20, and 30 days
  Total phospholipid concentration
  Individual phospholipid concentration (lyso phosphatidylcholine, phosphatidylcholine, sphingomyelin, phosphatidylethanolamine, phosphatidylinositol)

SECONDARY OUTCOMES:
Plasma lipids | after 0,10,20, and 30 days
  Fatty acid fraction (total fatty acid distribution, phospholipid fatty acid distribution)
  Cholesterol fraction (total cholesterol, LDL cholesterol, HDL cholesterol)
  Triacylglycerides fraction
Fecal lipids | after 0,10,20, and 30 days
  Fecal lipids (crude fat, total phospholipids, sterols, bile acids)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller University, Department of Nutritional Physiology
Locations (1):
- Friedrich Schiller University of Jena, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Keller S, Malarski A, Reuther C, Kertscher R, Kiehntopf M, Jahreis G. Milk phospholipid and plant sterol-dependent modulation of plasma lipids in healthy volunteers. Eur J Nutr. 2013 Apr;52(3):1169-79. doi: 10.1007/s00394-012-0427-0. Epub 2012 Jul 27. PMID 22836514